CLINICAL TRIAL: NCT02702466
Title: Evaluation of the Effectiveness of Personalized Short and Intensive Educational SPA Therapy Prevention of Upper Limb Musculoskeletal Disorders (MSDs).
Brief Title: Active Prevention of Upper Limb Musculoskeletal Disorders in Thermal Environment (MUSKA).
Acronym: MUSKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUSKA
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Musculoskeletal Disorders
Keywords: Upper limb musculoskeletal disorders; Spa treatment; Randomized controlled trials; Education; Self- management; Self-care; Exercise; Non pharmacological treatment
MeSH Terms: conditions — Musculoskeletal Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate SPA Therapy (Experimental): 6 day immediate SPA treatment (soon after randomization) and written information with physical exercises adapted to their pathology and also a program of healthcare at the USB key
  Interventions: Other: SPA Therapy
- Late SPA Therapy (Active Comparator): Written information with physical exercises adapted to their pathology and a program of healthcare at the USB key and late 6 day SPA treatment
  Interventions: Other: SPA Therapy

INTERVENTIONS:
Other: SPA Therapy — Immersion bath and shower ( 1 treatment ) Underwater shower with localized massage on the painful area ( 1 treatment ) or equivalent underwater massage Illutations ( 1 treatment ) or equivalent ( poultice ) Mobilization Pool ( 1 care) Education to exercise
  Other Names: Non pharmacological intervention

SUMMARY:
The main objective of this work is to demonstrate superiority to three months of a standardized short course of SPA Therapy of 6 days associated with personalized health education program compared to conventional therapy in the management of MSDs on the functional capabilities of the employees in their daily lives (personal or professional)

DETAILED DESCRIPTION:
Musculoskeletal disorders are the leading occupational disease in industrialized countries. The symptoms are varied, their multiple risk factors, work organization may be involved. Musculoskeletal disorders affect the muscles, tendons and nerves of the mainly upper limbs (neck, shoulder, elbow, wrist and hand). Pain or functional impairment are common to all these disorders.The proposed study is part of an active preventive approach in addressing current employees with latent or symptomatic upper extremity MSD linked to a hyper solicitation. This study provide them 6 days SPA therapy (before or after work) combined with a health education program to help improve their lives over time.

ELIGIBILITY:
Inclusion Criteria:

* TMS latent or symptomatic of the upper limbs according to the European Consensus SALTSA / Q score with INRS Nordic > 2
* With or without a history of work stoppage and occupation at the time of inclusion
* Age: > 18 years < 65 years
* Patient affiliated to a social security scheme ( beneficiary entitled )
* Patient has given its consent in writing to participate in the study

Exclusion Criteria:

* Contraindication to the spa therapy
* Spa achieved in the last 12 months
* Trouble behavior or understanding making it impossible to assess

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09; Primary Completion 2018-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The score from the scale Quick DASH | Month 03
  Change from baseline in measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb by Quick DASH measure

SECONDARY OUTCOMES:
Change of Quick DASH | Day 06, Month 01, Month 02, Month 03, Month 04, Month 05, Month 06
  Average change from baseline in measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb by Quick DASH measure
Pain intensity | Day 06, Month 01, Month 02, Month 03, Month 04, Month 05, Month 06
  Pain intensity measured on a Visual Analogical Scale (VAS)
Life quality | Day 06, Month 01, Month 02, Month 03, Month 04, Month 05, Month 06
  Life quality measured by SF36 (36-item Medical Outcomes Study Short-Form Health Survey - SF-36) Survey - SF-36)
Stopping time of work | Month 06
  Stopping time of work by self-administered questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (5):
- France (5):
  - Etablissement thermal, Aix-les-Bains, Auvergne-Rhône-Alpes
  - Etablissement thermal, Châtel-Guyon, Auvergne-Rhône-Alpes
  - Etablissement thermal, Royat, Auvergne-Rhône-Alpes
  - Etablissement thermal, Saint-Amand-les-Eaux, Hauts-de-France
  - Etablissement thermal, Balaruc-les-Bains, Occitanie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McBeth J, Jones K. Epidemiology of chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):403-25. doi: 10.1016/j.berh.2007.03.003. PMID 17602991
- [Background] Kamaleri Y, Natvig B, Ihlebaek CM, Bruusgaard D. Localized or widespread musculoskeletal pain: does it matter? Pain. 2008 Aug 15;138(1):41-46. doi: 10.1016/j.pain.2007.11.002. Epub 2008 Feb 20. PMID 18077092
- [Background] Solidaki E, Chatzi L, Bitsios P, Markatzi I, Plana E, Castro F, Palmer K, Coggon D, Kogevinas M. Work-related and psychological determinants of multisite musculoskeletal pain. Scand J Work Environ Health. 2010 Jan;36(1):54-61. doi: 10.5271/sjweh.2884. Epub 2009 Dec 11. PMID 20011982
- [Background] Fan ZJ, Smith CK, Silverstein BA. Assessing validity of the QuickDASH and SF-12 as surveillance tools among workers with neck or upper extremity musculoskeletal disorders. J Hand Ther. 2008 Oct-Dec;21(4):354-65. doi: 10.1197/j.jht.2008.02.001. PMID 19006762
- [Background] Polson K, Reid D, McNair PJ, Larmer P. Responsiveness, minimal importance difference and minimal detectable change scores of the shortened disability arm shoulder hand (QuickDASH) questionnaire. Man Ther. 2010 Aug;15(4):404-7. doi: 10.1016/j.math.2010.03.008. PMID 20434942
- [Background] Fayad F, Lefevre-Colau MM, Gautheron V, Mace Y, Fermanian J, Mayoux-Benhamou A, Roren A, Rannou F, Roby-Brami A, Revel M, Poiraudeau S. Reliability, validity and responsiveness of the French version of the questionnaire Quick Disability of the Arm, Shoulder and Hand in shoulder disorders. Man Ther. 2009 Apr;14(2):206-12. doi: 10.1016/j.math.2008.01.013. Epub 2008 Apr 23. PMID 18436467
- [Background] Fayad F, Lefevre-Colau MM, Mace Y, Fermanian J, Mayoux-Benhamou A, Roren A, Rannou F, Roby-Brami A, Gautheron V, Revel M, Poiraudeau S. Validation of the French version of the Disability of the Arm, Shoulder and Hand questionnaire (F-DASH). Joint Bone Spine. 2008 Mar;75(2):195-200. doi: 10.1016/j.jbspin.2007.04.023. Epub 2007 Aug 30. PMID 17983829
- [Result] Meroni R, Scelsi M, Boria P, Sansone V. Shoulder disorders in female working-age population: a cross sectional study. BMC Musculoskelet Disord. 2014 Apr 4;15:118. doi: 10.1186/1471-2474-15-118. PMID 24708552
- [Result] Parot-Schinkel E, Descatha A, Ha C, Petit A, Leclerc A, Roquelaure Y. Prevalence of multisite musculoskeletal symptoms: a French cross-sectional working population-based study. BMC Musculoskelet Disord. 2012 Jul 20;13:122. doi: 10.1186/1471-2474-13-122. PMID 22818516
- [Derived] Lanhers C, Grolier M, Dutheil F, Gay C, Goldstein A, Mourgues C, Levyckyj C, Pereira B, Coudeyre E. Comparison of self-management and spa therapy for upper-extremity musculoskeletal disorders: A randomized controlled trial. Ann Phys Rehabil Med. 2024 Apr;67(3):101813. doi: 10.1016/j.rehab.2023.101813. Epub 2024 Mar 12. PMID 38479114
- [Derived] Lanhers C, Pereira B, Gay C, Herisson C, Levyckyj C, Dupeyron A, Coudeyre E. Evaluation of the efficacy of a short-course, personalized self-management and intensive spa therapy intervention as active prevention of musculoskeletal disorders of the upper extremities (Muska): a research protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2016 Dec 9;17(1):497. doi: 10.1186/s12891-016-1353-8. PMID 27938361